CLINICAL TRIAL: NCT05806970
Title: Email Nudges to Improve GDMT (MRA) Adherence in Heart Failure
Acronym: ENIGMA-HF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Converted clinical trial approach to a quality improvement approach
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Nicholas K. Brownell, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UCLA IRB#23-000305
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Ambulatory Care; Learning Health System; Quality Improvement [QI]; Implementation Science; Clinical Decision Support; Mineralocorticoid Receptor Antagonist [MRA]; Guideline Directed Medical Therapy [GDMT]

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Email Nudge (Experimental): The intervention will include contacting UCLA Health Cardiology clinic managers with a list of all HFrEF patients eligible for an MRA who are cared for by a provider randomized to the intervention arm. Clinic managers will be asked to make an appointment in the next 60 days for these patients with the specific indication: GDMT initiation - consider MRA. If an appointment is already present in the next 60 days, the indication will be changed to: GDMT initiation - consider MRA.
  Interventions: Other: Email Nudge
- No Intervention - Control Group (No Intervention): Providers randomized to the control arm will perform clinical duties as usual. Their patients will receive routine clinical care.

INTERVENTIONS:
Other: Email Nudge — An email to UCLA Health Cardiology clinic managers with a list of MRA-eligible HFrEF patients and a request to schedule or change cardiology appointments.
  Arms: Intervention - Email Nudge

SUMMARY:
The Email Nudges to Improve GDMT (MRA) Adherence in Heart Failure (ENIGMA-HF) study is a pragmatic parallel-arm randomized control trial of a quality improvement (QI) intervention involving email nudges to cardiology clinic managers to schedule appointments specific to guideline directed medical therapy (GDMT) initiation, with the goal of optimizing mineralocorticoid-receptor antagonist (MRA) use by patients with heart failure with reduced ejection fraction (HFrEF) cared for by cardiologists within the University of California, Los Angeles (UCLA) Health System.

DETAILED DESCRIPTION:
Importance: Guideline directed medical therapy (GDMT) is a specific set of 4 medications proven to improve morbidity and mortality for patients with heart failure (HF) with reduced ejection fraction (HFrEF), yet they are underutilized nationally and internationally. Various quality improvement (QI) interventions have had varying degrees of success at increasing GDMT prescription and titration.

Objective: The purpose of the study is to assess whether email nudges to UCLA Health cardiology clinic managers to schedule GDMT-specific appointments can lead to increased utilization of a specific medication within GDMT called a mineralocorticoid-receptor antagonist (MRA). Pertinent secondary objectives will include evaluating whether email nudges specific to MRA would increase utilization of the other medications in GDMT and whether they would increase appointments specific to GDMT.

Design, Setting, and Participants: The basic design is a pragmatic parallel-arm randomized control trial of a QI intervention. The setting is cardiology outpatient clinics at a large university-based single integrated healthcare system (UCLA Health). Participants are outpatients with HFrEF under the care of a UCLA cardiologist, with an ejection fraction on file, and currently not prescribed an MRA.

Hypothesis: The investigators hypothesize that the intervention will lead to an increased utilization of MRA, compared to the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Facility: UCLA Health System
* Patient is 18 years of age or older
* Patient is under the care of a UCLA cardiologist
* Patient has a primary diagnosis of HFrEF
* Patient is not currently prescribed an MRA

Exclusion Criteria:

* Hyperkalemia
* Chronic kidney disease stage 4 or higher
* Pregnant or breastfeeding patients
* Heart transplant or ventricular-assist device patients
* Hospice patients
* Patients without an LVEF on file
* Patients with an EF >35%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of eligible patients prescribed MRA | 60 days
  Proportion of patients that receive an active prescription for mineralocorticoid receptor antagonist (MRA) compared between arms at the end of the study.

SECONDARY OUTCOMES:
Percentage of eligible patients prescribed ACE/ARB/ARNI, beta blocker, or SGLT2i | 60 days
  Proportion of patients that receive an active prescription for angiotensin-converting enzyme inhibitor (ACE), angiotensin II receptor blocker (ARB), angiotensin receptor neprilysin inhibitor (ARNI), beta blocker, or sodium-glucose cotransporter-2 inhibitor (SGLT2i) compared between arms at the end of the study.
Percentage of eligible patients prescribed ACE/ARB/ARNI | 60 days
  Proportion of patients that receive an active prescription for angiotensin-converting enzyme inhibitor (ACE), angiotensin II receptor blocker (ARB), or angiotensin receptor neprilysin inhibitor (ARNI) compared between arms at the end of the study.
Percentage of eligible patients prescribed ARNI | 60 days
  Proportion of patients that receive an active prescription for angiotensin receptor neprilysin inhibitor (ARNI) compared between arms at the end of the study.
Percentage of eligible patients prescribed beta blocker | 60 days
  Proportion of patients that receive an active prescription for beta-blocker compared between arms at the end of the study.
Percentage of eligible patients prescribed SGLT2i | 60 days
  Proportion of patients that receive an active prescription for sodium-glucose cotransporter-2 inhibitor (SGLT2i) compared between arms at the end of the study.

OTHER OUTCOMES:
Percentage of eligible patients who have an appointment scheduled or indication changed in 60 days | 60 days
  Proportion of patients that have an appointment actively scheduled or an appointment indication actively changed within 60 days of study initiation.
Percentage of eligible patients who have an appointment scheduled in 60 days | 60 days
  Proportion of patients that have an appointment actively scheduled within 60 days of study initiation.
Percentage of eligible patients who have an appointment indication changed in 60 days | 60 days
  Proportion of patients that have an appointment already scheduled within 60 days of study initiation, but have the indication changed to "GDMT initiation - consider MRA."
Percentage of eligible patients who have a BMP ordered after MRA initiation | 60 days
  Safety endpoint: Proportion of patients that receive an active order for a basic metabolic panel (BMP) after being prescribed a mineralocorticoid receptor antagonist (MRA)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas K Brownell, MD, Principal Investigator — University of California, Los Angeles; David J Cho, MD MBA, Principal Investigator — University of California, Los Angeles; Pooya I Bokhoor, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brownell NK, Ziaeian B, Fonarow GC. The Gap to Fill: Rationale for Rapid Initiation and Optimal Titration of Comprehensive Disease-modifying Medical Therapy for Heart Failure with Reduced Ejection Fraction. Card Fail Rev. 2021 Nov 26;7:e18. doi: 10.15420/cfr.2021.18. eCollection 2021 Mar. PMID 34950508